CLINICAL TRIAL: NCT00557687
Title: Prediction of Ovarian Response After Ovarian Stimulation for in Vitro Fertilization
Brief Title: Prediction of Ovarian Response
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor, Aristotle University Of Thessaloniki
Other Study IDs: UHR-5
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: In Vitro Fertilization
Keywords: IVF; ovarian reserve; poor response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum

SUMMARY:
The purpose of this study is to evaluate if there is an association between the endocrine and ultrasonographic markers of ovarian reserve and the IVF outcome and to determine which markers contribute to the prediction of poor response in IVF.

DETAILED DESCRIPTION:
One of the most frustrating problem in IVF today is that of poor ovarian response. There is an amount of woman undergoing infertility treatment, who respond poorly to the usual gonatotrophin stimulation protocol applied. The ovarian response, which is the number of antral follicles and oocytes which are developed in the ovary after stimulation, is correlated directly with the ovarian reserve. As ovarian reserve is defined the existent quantitative and qualitative supply of follicles which are found in the ovaries and potentially can be developed in dominant and therefore it is closely associated with reproductive potential.

There is a plethora of criteria used to characterize the poor response. The number of developed follicles or the number of oocytes retrieved after a standard dose ovarian stimulation protocol, are two of the most substantial criteria for the definition of poor ovarian reserve. Satisfying response after ovulation induction is considered the retrieval of 5-14 oocytes per patient, whereas poor response is considered the retrieval of 4 or less oocytes. Using the standard doses, however, a number of patients will exhibit inappropriate ovarian responses. Exaggerated response leads to increased risk of ovarian hyperstimulation syndrome, while on the other hand, inadequate ovarian response is associated with increased number of IVF cancellations.

During the past two decades, a substantial amount of research has been carried out in order to improve our knowledge on ovarian response predictors. Age has often guided infertility treatment choices, since a woman's chronological age is the single most important factor in predicting a couple's reproductive potential, as it is generally acknowledged that reproductive ageing is related to both quantitative and qualitative reduction of the primordial follicle pool. However, age alone is of limited value and so it cannot predict the response to infertility treatment.

A number of ovarian reserve tests have been designed in order to determine ovarian reserve and have been evaluated for their ability to predict the outcome of IVF. Many of these tests have become part of the routine diagnostic procedure for infertile patients who undergo assisted reproductive techniques. These ovarian reserve tests include the measurement of specific endocrine markers in combination with the study of some ultra-sonographic parameters.

Basal FSH was the first widely used endocrine marker of ovarian reserve that had better potential than age for predicting decreased ovarian function and today it is established that patients with elevated basal FSH levels have lowered success rates after IVF. At present, several other markers of ovarian reserve are advocated, such as basal estradiol levels, basal LH levels, early follicular phase serum inhibin B concentration and anti-mullerian hormone concentration.

Moreover, several ovarian ultrasonographic parameters are studied as markers for ovarian resposiveness. The antral follicle count, the ovarian volume and the ovarian stromal blood flow appeared to be indicative of poor response in assisted reproduction.

The purpose of this prospective study is to evaluate if there is an association between the endocrine and ultrasonographic markers of ovarian reserve and the IVF outcome and to determine which markers contribute to the prediction of poor response in IVF.

ELIGIBILITY:
Inclusion Criteria:

* Age < 39 years
* Presence of both ovaries
* FSH levels < 12,5 IU/l
* Duration of mensrual cycle >21 days and <35days

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing ovarian stimulation with gonadotropins and GnRH antagonists for IVF
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
prediction of poor ovarian response | at oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Basil C Tarlatzis, Study Director — Unit for Human Reproduction, 1st Dept of Obstetrics and Gynaecology
Locations (1):
- Unit for Human Reproduction, Thessaloniki, Greece